CLINICAL TRIAL: NCT02633943
Title: Long-term Follow-up of Subjects With Transfusion-Dependent β-Thalassemia (TDT) Treated With Ex Vivo Gene Therapy Using Autologous Hematopoietic Stem Cells Transduced With a Lentiviral Vector
Brief Title: Long-term Follow-up of Subjects With Transfusion-Dependent β-Thalassemia (TDT) Treated With Ex Vivo Gene Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LTF-303
Record Dates: First submitted 2015-11-30; First posted 2015-12-17 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Transfusion-dependent Beta-Thalassemia
MeSH Terms: interventions — Safety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with Transfusion-Dependent β-Thalassemia: Long-term follow-up for participants treated with ex vivo gene therapy product in applicable bluebird bio-sponsored parent clinical trials and who agreed to participate in this study. Participants will be followed in this study for 13 years (for a total of 15 years of follow-up after drug product infusion in the parent studies)
  Interventions: Other: Safety and efficacy assessments

INTERVENTIONS:
Other: Safety and efficacy assessments — Genetic: No interventional drug product utilized in this follow-up study
  Participants received a single IV infusion of LentiGlobin BB305 Drug Product in the parent studies. Vector copy number (VCN) measurement, safety evaluations, disease-specific assessments, and assessments to monitor for long-term effects of autologous transplant are conducted in this study.

SUMMARY:
This is a multi-center, long-term safety and efficacy follow-up study for subjects with transfusion-dependent β-thalassemia (TDT) who have been treated with ex vivo gene therapy drug product in bluebird bio-sponsored parent clinical studies. After completing the parent clinical studies (approximately 2 years), eligible subjects will be followed for an additional 13 years for a total of 15 years post-drug product infusion. No investigational drug product will be administered in this study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent for this study by subjects, or as applicable, subject's parent(s)/legal guardian(s)
* Treated with drug product for therapy of transfusion-dependent β-thalassemia in a bluebird bio-sponsored clinical study

Exclusion Criteria:

* There are no exclusion criteria for this study

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with transfusion-dependent β-thalassemia who have been treated with ex vivo gene therapy product in bluebird bio-sponsored clinical studies
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2035-11 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with malignancies | Up to 15 years post-drug product infusion
The number of subjects with immune-related AEs | Up to 15 years post-drug product infusion
The number of subjects with new or worsening hematologic disorders | Up to 15 years post-drug product infusion
The number of subjects with new or worsening neurologic disorders | Up to 15 years post-drug product infusion

SECONDARY OUTCOMES:
βA-T87Q-globin expression | Up to 15 years post-drug product infusion
  Median (min, max) βA-T87Q-globin expression
Proportion of subjects treated with beti-cel who achieved Transfusion Independence (TI) | Up to 15 years post-drug product infusion
  Proportion of subjects who achieved TI, defined as a weighted average Hb ≥ 9 g/dL without any packed red blood cell (pRBC) transfusions for a continuous period of ≥ 12 months at any time after drug product infusion in parent study and/or Study LTF-303
Proportion of subjects treated with beti-cel who achieved Transfusion Independence at yearly timepoints | Up to 15 years post-drug product infusion
  Proportion of subjects treated with beti-cel who achieved TI at yearly timepoints including Year 5, Year 10, and Year 15 post-drug product infusion, and at last follow-up
Time from drug product infusion to achievement of Transfusion Independence (in parent study or Study LTF-303) | Up to 15 years post-drug product infusion
Duration of Transfusion Independence | Up to 15 years post-drug product infusion
Weighted average Hb during Transfusion Independence | Up to 15 years post-drug product infusion
Change in annualized pRBC transfusion volume (among subjects who achieved TI), from 6 months post-drug product infusion (parent study) through last follow-up | Up to 15 years post-drug product infusion
  Reduction in annualized pRBC transfusion volume (mL/kg/year) from 6 months post-drug product infusion (parent study) through last follow-up of at least 50%, 60%, 75%, 90%, or 100% as compared to the annualized pRBC transfusion volume during the 2 years prior to parent study enrollment
Annualized pRBC transfusion volume, from 6 months post-drug product infusion (parent study) through last follow-up | Up to 15 years post-drug product infusion
  Annualized pRBC transfusion volume (mL/kg/year from 6 months post-drug product infusion (parent study) through last follow-up as compared to the annualized pRBC transfusion requirements during the 2 years prior to parent study enrollment
pRBC transfusion frequency, from 6 months post-drug product infusion (parent study) through last follow-up | Up to 15 years post-drug product infusion
  Annualized pRBC frequency (number/year) from 6 months post-drug product infusion (parent study) through last follow-up as compared to the annualized pRBC transfusion requirements during the 2 years prior to parent study enrollment
Time from drug product infusion to last pRBC transfusion (in parent study or Study LTF-303) | Up to 15 years post-drug product infusion
Time from last pRBC transfusion (in parent study or Study LTF-303) to last follow-up | Up to 15 years post-drug product infusion
Weighted average nadir Hb from 6 months post-drug product infusion (parent study) through last follow-up | Up to 15 years post-drug product infusion
  Weighted average nadir Hb from 6 months post-drug product infusion (parent study) through last follow-up as compared to the weighted average nadir Hb during the 2 years prior to parent study enrollment
Unsupported total Hb levels over time through last follow-up | Up to 15 years post-drug product infusion
  Unsupported total Hb level is defined as the total Hb measurement level without any acute or chronic pRBC transfusions within 60 days prior to the measurement date.
Proportion of subjects with unsupported total Hb levels ≥ 10 g/dL over time through last follow-up, including Year 5, Year 10, and Year 15 | Up to 15 years post-drug product infusion
Proportion of subjects with unsupported total Hb levels ≥ 11 g/dL over time through last follow-up, including Year 5, Year 10, and Year 15 | Up to 15 years post-drug product infusion
Proportion of subjects with unsupported total Hb levels ≥ 12 g/dL over time through last follow-up, including Year 5, Year 10, and Year 15 | Up to 15 years post-drug product infusion
Proportion of subjects with unsupported total Hb levels ≥ 13 g/dL over time through last follow-up, including Year 5, Year 10, and Year 15 | Up to 15 years post-drug product infusion
Proportion of subjects with unsupported total Hb levels ≥ 14 g/dL over time through last follow-up, including Year 5, Year 10, and Year 15 | Up to 15 years post-drug product infusion
Liver iron content (LIC) by magnetic resonance imaging (MRI)/Superconducting Quantum Interference Device (SQUID) over time at yearly timepoints through last follow-up | Up to 15 years post-drug product infusion
Change from parent study baseline in LIC by MRI/SQUID over time at yearly timepoints through last follow-up | Up to 15 years post-drug product infusion
Cardiac T2* by MRI over time at yearly timepoints through last follow-up | Up to 15 years post-drug product infusion
Change from parent study baseline in cardiac T2* by MRI over time at yearly timepoints through last follow-up | Up to 15 years post-drug product infusion
Serum ferritin over time at yearly timepoints through last follow-up | Up to 15 years post-drug product infusion
Change from parent study baseline in serum ferritin over time at yearly timepoints through last follow-up | Up to 15 years post-drug product infusion
Number of subjects who stopped iron chelation post-DP infusion | Up to 15 years post-drug product infusion
  Defined as subjects who stopped iron chelation or never restarted chelation after DP infusion.
Number of subjects who stopped iron chelation for at least 6 months post-drug product infusion | Up to 15 years post-drug product infusion
Time from stopping chelation to last follow-up | Up to 15 years post-drug product infusion
  Among subjects that never restart chelation after DP infusion.
Proportion of subjects using phlebotomy therapy post-drug product infusion | Up to 15 years post-drug product infusion
Annualized frequency of phlebotomy therapy usage | Up to 15 years post-drug product infusion
  Annualized frequency of phlebotomy therapy usage is defined as the number of procedures per year, calculated from DP infusion through last follow-up.
Reticulocyte counts over time at yearly timepoints through last follow-up | Up to 15 years post-drug product infusion
Change from Baseline in reticulocyte counts at yearly timepoints through last follow-up | 15 years post-drug product infusion
  Baseline defined as value closest, but prior to, conditioning in parent study.
Proportion of subject with nucleated RBC over time at yearly timepoints through last follow-up | Up to 15 years post-drug product infusion
Change from Baseline in patient reported outcome (PRO) as assessed by Pediatric Quality of Life Inventory (PedsQL | 5 years post-drug product infusion
Change from Baseline in PRO as assessed by EuroQol-5D Youth version (EQ-5D-Y) | 5 years post-drug product infusion
Change from Baseline in PRO as assessed by EuroQol-5D (EQ-5D-3L) | 5 years post-drug product infusion
Change From Baseline in PRO as assessed by Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) Questionnaire Score | 5 years post-drug product infusion
Change from Baseline in PRO as assessed by Short Form-36 Health Survey (SF-36) | 5 years post-drug product infusion

CONTACTS AND LOCATIONS:
Overall Officials: Himal L Thakar, MD, Study Director — bluebird bio, Inc.
Locations (15):
- United States (6):
  - Oakland, California
  - Chicago, Illinois
  - Bethesda, Maryland
  - New York, New York
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
- Sydney, Australia
- France (2):
  - Marseille
  - Paris
- Germany (2):
  - Hanover
  - Heidelberg
- Thessaloniki, Greece
- Rome, Italy
- Bangkok, Thailand
- London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Bluebird bio is committed to transparency and appropriately de-identified subject-level datasets and supporting documents may be shared after all participants have completed study participation and following attainment of applicable marketing approvals associated with a given study and consistent with criteria established by bluebird bio and/or industry best practices to maintain the privacy of study participants. For enquiries, please contact us at datasharing@bluebirdbio.com.

REFERENCES:
- [Derived] Kwiatkowski JL, Thompson AA, Schneiderman J, Thuret I, Kulozik AE, Yannaki E, Cavazzana M, Hongeng S, Olson TS, Sauer MG, Thrasher AJ, Lal A, Rasko JE, Kunz JB, Kinney MA, Chawla A, Ali S, Tao G, Thakar H, Paramore C, Witthuhn N, Walters MC, Locatelli F. Long-term efficacy and safety results of betibeglogene autotemcel gene therapy for transfusion-dependent beta-thalassemia. Blood. 2026 Jan 12:blood.2025029196. doi: 10.1182/blood.2025029196. Online ahead of print. PMID 41525466
- [Derived] Kwiatkowski JL, Walters MC, Hongeng S, Yannaki E, Kulozik AE, Kunz JB, Sauer MG, Thrasher AJ, Thuret I, Lal A, Tao G, Ali S, Thakar HL, Elliot H, Lodaya A, Lee J, Colvin RA, Locatelli F, Thompson AA. Betibeglogene autotemcel gene therapy in patients with transfusion-dependent, severe genotype beta-thalassaemia (HGB-212): a non-randomised, multicentre, single-arm, open-label, single-dose, phase 3 trial. Lancet. 2024 Nov 30;404(10468):2175-2186. doi: 10.1016/S0140-6736(24)01884-1. Epub 2024 Nov 8. PMID 39527960
- [Derived] Magrin E, Semeraro M, Hebert N, Joseph L, Magnani A, Chalumeau A, Gabrion A, Roudaut C, Marouene J, Lefrere F, Diana JS, Denis A, Neven B, Funck-Brentano I, Negre O, Renolleau S, Brousse V, Kiger L, Touzot F, Poirot C, Bourget P, El Nemer W, Blanche S, Treluyer JM, Asmal M, Walls C, Beuzard Y, Schmidt M, Hacein-Bey-Abina S, Asnafi V, Guichard I, Poiree M, Monpoux F, Touraine P, Brouzes C, de Montalembert M, Payen E, Six E, Ribeil JA, Miccio A, Bartolucci P, Leboulch P, Cavazzana M. Long-term outcomes of lentiviral gene therapy for the beta-hemoglobinopathies: the HGB-205 trial. Nat Med. 2022 Jan;28(1):81-88. doi: 10.1038/s41591-021-01650-w. Epub 2022 Jan 24. PMID 35075288
- See also: HGB-204 Clinicaltrials.gov — https://www.clinicaltrials.gov/ct2/show/NCT01745120?term=lentiglobin&rank=2
- See also: HGB-205 Clinicaltrials.gov — https://www.clinicaltrials.gov/ct2/show/NCT02151526?term=lentiglobin&rank=3
- See also: HGB-207 Clinicaltrials.gov — https://clinicaltrials.gov/ct2/show/NCT02906202
- See also: HGB-212 Clinicaltrials.gov — https://clinicaltrials.gov/ct2/show/NCT03207009?term=HGB-212&recrs=a&rank=1